CLINICAL TRIAL: NCT00846274
Title: Single-Dose, Open Label, Randomized Comparative Clinical Trial to Evaluate the Tolerability, Safety and PK/PD of Human ATIII Products, "SKATIII Injection" and"ATIII Injection" in Healthy Male Subjects
Brief Title: Phase1 Syudy to Evaluate the Safety and PK/PD of Human Antithrombin III
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SK Chemicals Co., Ltd. (Industry)
Collaborators: Korea University Anam Hospital (Other)
Responsible Party: Clinical Research Team, SK Chemicals Co.,Ltd.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SKATIII_I_2007
Record Dates: First submitted 2009-02-16; First posted 2009-02-18 (Estimated); Last update posted 2009-02-18 (Estimated); Status verified 2009-02

CONDITIONS: Healthy
Keywords: Healthy Male subjects

ARMS (2):
- Antithrombin III (Active Comparator)
  Interventions: Biological: SK Antithrombin III
- SK Antithrombin III (Experimental)
  Interventions: Biological: SK Antithrombin III

INTERVENTIONS:
Biological: SK Antithrombin III

SUMMARY:
To evaluate the PK/PD of single injected human ATIII Products, SKATIII and ATIII, phase1 study in healthy male subjects was designed

ELIGIBILITY:
Inclusion Criteria:

* ages 19 to 40
* Body weight: More than 50kg
* Healthy male subject

Exclusion Criteria:

* Hb<14g/dL, Hct<42%
* ATIII hypersensitivity

Ages: 19 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-10; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
ATIII activity | within 20min after injection ATIII

SECONDARY OUTCOMES:
ATIII antigen | within 20min after injection ATIII

CONTACTS AND LOCATIONS:
Overall Officials: Ji Young Park, MD,PhD, Principal Investigator — Korea University Anam Hospital
Locations (1):
- SK chemicals, Seoul, South Korea

REFERENCES:
- [Derived] Kim KA, Lim YY, Kim SH, Park JY. Bioequivalence of two intravenous formulations of antithrombin III: a two-way crossover study in healthy Korean subjects. Clin Ther. 2013 Nov;35(11):1752-61. doi: 10.1016/j.clinthera.2013.08.018. Epub 2013 Oct 1. PMID 24094463